CLINICAL TRIAL: NCT05968261
Title: Implementation and Measurement of a Real-time, Near-remote Method to Operationalize Ultrasound-based Regional Anesthesia/Analgesia Procedural Techniques
Brief Title: Near Remote Method to Guide Performance of Regional Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Dr. Glenio Mizubuti (MD, PhD) (Other)
Responsible Party: Sponsor-Investigator, Dr. Glenio Mizubuti (MD, PhD), (MD, MSc, FRCPC, Associate Professor), Queen's University
Organization: Queen's University (Other)
Other Study IDs: 6038020
Record Dates: First submitted 2023-07-11; First posted 2023-08-01 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Analgesia; Nerve Block; Delivery of Healthcare; Hospitals, Teaching
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Real time 'near remote' guidance of regional blocks — Trainees who are to perform regional blocks will do so under expert guidance via tele-mentoring. This will be done using a novel technology consisting of a wirelessly linked iPad which will display the ultrasound image to the block operator/trainee. This image will be concurrently visualized by an expert mentor through their smartphone, who will then provide feedback/guidance in real-time to the operator/trainee.

SUMMARY:
Ultrasound-guided regional anesthesia/analgesia techniques (or simply, 'regional blocks') have gained popularity as they can reduce, and sometimes even eliminate, the need for opiate analgesics (and, consequently, their side effects), thereby improving patient safety, reducing length of hospital stay and medical costs, and improving patient satisfaction. However, a major barrier to mainstream uptake of such techniques relates to training. These techniques require the acquisition of new skills under expert guidance, which is often not possible given the daily demands placed upon anesthesiologists. As a result, many opportunities for providing regional blocks may be missed.

The purpose of this study is to implement a new real-time 'near remote' guidance method in which trainees who are to perform regional blocks can do so via tele-mentoring under expert guidance. This will be done using a novel technology whereby the ultrasound image is concurrently displayed on an iPad screen (for the block operator/trainee) as well as on the (near remotely supervising) expert mentor's smartphone. Trainees and mentors will use this method to perform various standard of care regional blocks, either in the perioperative or emergency department settings. Participants' opinions of the novel teaching and learning method will be assessed.

DETAILED DESCRIPTION:
Ultrasound-guided regional anesthesia/analgesia techniques (herein referred to simply as 'regional blocks') have gained popularity as they can reduce, and sometimes even eliminate, the need for opiate analgesics (and, consequently, their side effects), thereby improving patient safety, reducing length of hospital stay and medical costs, and improving patient satisfaction. However, a major barrier to mainstream uptake of such techniques relates to training. These techniques require the acquisition of new skills under expert guidance, which is often not possible given the daily time-sensitive and competing demands placed upon anesthesiologists. Furthermore, staff shortages and increasing demands caused by the COVID-19 pandemic have limited expert availability for one-on-one guidance even more. As a result, many opportunities for providing regional analgesia may be missed or performed in the absence of expert guidance.

Currently, expert staff regional anesthesiologists would ideally be available to supervise regional blocks. In clinical practice, however, if no staff regional anesthesiologist is available to supervise, senior anesthesia residents (post-graduate years 3 to 5) will often proceed with performing lower-risk blocks (e.g., adductor canal blocks) independently provided they feel confident and comfortable with the technique. If, however, the senior anesthesia resident is not comfortable with performing a higher-risk block without supervision, the patient would likely then receive general anesthesia combined with a multimodal analgesic regimen for perioperative pain control.

The purpose of the current study is to implement a new real-time 'near-remote' guidance method, in which trainees who are to perform regional blocks can do so via tele-mentoring under expert guidance. This will be done using an ultrasound-linked iPad which is a novel technology whereby the high-resolution ultrasound image is concurrently displayed on an iPad screen (for the block operator/trainee) as well as on the (near remotely supervising) expert mentor's smartphone. The expert mentor will either be at a distance in the same room or in an adjacent room, but readily available to intervene quickly if necessary. Trainees and mentors will use this method to perform various standard of care regional blocks on patients, either prior to elective surgical procedures or in the emergency department in the context of trauma injuries. All regional blocks will be as per standard of care, except they will be performed under expert 'near-remote' guidance.

Following the regional block performed via tele-mentored expert-guidance, both the trainee and mentor will complete a questionnaire pertaining to that particular block. Questionnaires will be completed electronically via Qualtrics. Block success will also be assessed (i.e., sensory block to ice within 30 min following block performance, as per standard of care) and documented. Towards the end of the study, voluntary focus group sessions will be held, during which trainees and mentors will have the opportunity to provide feedback regarding the newly implemented teaching and learning method. Thematic analyses will then be conducted.

Success with the current study may lay the groundwork for future research investigations to examine the feasibility of guiding such blocks by more remote methods (i.e., with the expert more than a few feet away).

ELIGIBILITY:
Inclusion Criteria:

* Mentors: Staff anesthesiologists who are experts in regional blocks.
* Trainees: Senior (PGY3-5) residents (anesthesiology and emergency medicine), and staff (emergency medicine) physicians who have already performed and are comfortable with being supervised near remotely for the regional block at hand.
* Patients: Greater or equal to 18 years of age presenting for surgery or with traumatic injuries amenable to regional blocks.
* All of the above: Able to read and understand English, and competent to provide written informed consent.

Exclusion Criteria:

* Mentors: Staff anesthesiologists who are not experts in the performance/teaching of regional blocks.
* Trainees: Junior (PGY1-2) residents (for any/all types of regional blocks), and senior (PGY3-5) residents and staff physicians who are not comfortable with being supervised near remotely for the regional block at hand.
* Patients: Less than 18 years of age.
* All of the above: Unable to read and understand English, and not competent to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include: (1) mentors, i.e., staff regional anesthesiologists who are experts in ultrasound-guided regional blocks; (2) trainees, i.e., PGY-3 to PGY-5 anesthesia and emergency medicine residents, and emergency medicine staff physicians; and (3) patients, i.e., individuals 18 years and older scheduled for surgery amenable to regional blocks or presenting to the emergency department with traumatic injuries amenable to regional blocks.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Participant opinion | Immediately following block performance
  The investigators will assess the opinions of mentors and trainees regarding the use of 'near-remote' guidance for the performance of ultrasound-guided regional blocks.

SECONDARY OUTCOMES:
Block success | Within 30 min following block performance
  Patients' sensation to ice
Block image | Through study completion, an average of 1 year
  Saved ultrasound image at the end of the block procedure. Specifically, this image will be saved after completion of local anesthetic injection and before removal of the block needle for subsequent review by a blinded expert.
Complications | Immediately postoperatively
  Any complications associated with performed regional blocks
Patient satisfaction | Immediately postoperatively
  Patient satisfaction with block performance
Number of attempts | Immediately following block performance
  Number of attempts to successfully perform regional block
Participant feedback | Through study completion, an average of 1 year
  Qualitative feedback from trainees and mentors via focus groups

CONTACTS AND LOCATIONS:
Overall Officials: Glenio B. Mizubuti, MD, MSc, FRCPC, Principal Investigator — Queen's University. Department of Anesthesiology and Perioperative Medicine
Locations (1):
- Hotel Dieu Hospital site (primary) and Kingston General Hospital site (secondary), Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
The information which will be associated (via study ID number) with each ultrasound image includes: sex, age, BMI range, surgery type and regional block type. The data will be saved directly to a secure server, and subsequently exported to SPSS for analysis. The only identifier will be the study ID number.

REFERENCES:
- See also: Exploring the utility of assistive artificial intelligence for ultrasound scanning in regional anesthesia — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9046753/
- See also: Regional anesthesia training model for resource-limited settings: a prospective single-center observational study with pre-post evaluations — https://pubmed.ncbi.nlm.nih.gov/32447288/
- See also: Application of distant live broadcast in clinical anesthesiology teaching — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8991162/
- See also: FaceTime® for teaching ultrasound-guided anesthetic procedures in remote place — https://pubmed.ncbi.nlm.nih.gov/24222344/
- See also: Novel real-time feedback and integrated simulation model for teaching and evaluating ultrasound-guided regional anesthesia skills in pediatric anesthesia trainees — https://pubmed.ncbi.nlm.nih.gov/22612411/